CLINICAL TRIAL: NCT06482502
Title: Investigation of the Validity and Reliability of the 6-Minute Pegboard and Ring Test in Parkinson's Patients for Upper Extremity Endurance Assessments
Brief Title: Validity of the 6-Minute Pegboard and Ring Test in Parkinson's Patients
Status: Recruiting | Type: Observational
Sponsor: Emre Şenocak (Other)
Responsible Party: Sponsor-Investigator, Emre Şenocak, Research Assisstant, Karadeniz Technical University
Organization: Karadeniz Technical University (Other)
Other Study IDs: 2024/77
Record Dates: First submitted 2024-06-26; First posted 2024-07-01 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson; Validity; 6-Minute Pegboard and Ring Test
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 6-MPRT Group: There is 1 group in the study. All assessments are made on the same group.

SUMMARY:
Tests used to assess upper extremity endurance in Parkinson's patients are limited. This study aimed to investigate whether the 6-Minute Pegboard and Ring Test (6-MPRT), which has been validated in many respiratory disease groups in previous studies, is an endurance assessment battery that can also be used in Parkinson's patients. 6-MPRT, Weight Lifting Test, and 30-Second Arm Curl Test will be applied in the assessments. Assessments will be made twice on the same day by two different evaluators, 1 hour apart. After the first evaluation, the patient will be called for the second time 2 days later, and the same procedure will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Hoehn & Yahr staging ≤3 points,
* Individuals who have not undergone a rehabilitation program of at least 20 days in the last 6 months,
* Those with full upper extremity shoulder flexion and abduction active joint range of motion.

Exclusion Criteria:

* Those with severe heart disease such as heart failure, cardiac arrhythmia, hypertension,
* People with any orthopedic problem that will affect the upper extremity,
* Having a secondary neurological disease diagnosis,
* Having vision impairment that may affect measurement methods (not corrected by glasses),
* Having a cognitive disease that may cause difficulty in following the researchers' commands,
* Those who had changes in their medical use during the test (dose increase/decrease, drug change

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson Disease
Sampling Method: Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
6-Minute Pegboard and Ring Test | Baseline of the study (Assessor 1)
  The patient is in a sitting position. Opposite the patient are 4 metal rods located on a wooden table. Two of them are at shoulder level and the other two are 20 cm above shoulder level. During the test, the patient is asked to take the light rings at shoulder level with both hands at the same time and place them on the bars above. The higher the total number of rings carried indicates increased endurance.
6-Minute Pegboard and Ring Test | 2 days after the baseline assessment (Assessor 1)
  The patient is in a sitting position. Opposite the patient are 4 metal rods located on a wooden table. Two of them are at shoulder level and the other two are 20 cm above shoulder level. During the test, the patient is asked to take the light rings at shoulder level with both hands at the same time and place them on the bars above. The higher the total number of rings carried indicates increased endurance.
6-Minute Pegboard and Ring Test | Baseline of the study (Assessor 2)
  The patient is in a sitting position. Opposite the patient are 4 metal rods located on a wooden table. Two of them are at shoulder level and the other two are 20 cm above shoulder level. During the test, the patient is asked to take the light rings at shoulder level with both hands at the same time and place them on the bars above. The higher the total number of rings carried indicates increased endurance.
6-Minute Pegboard and Ring Test | 2 days after the baseline assessment (Assessor 2)
  The patient is in a sitting position. Opposite the patient are 4 metal rods located on a wooden table. Two of them are at shoulder level and the other two are 20 cm above shoulder level. During the test, the patient is asked to take the light rings at shoulder level with both hands at the same time and place them on the bars above. The higher the total number of rings carried indicates increased endurance.
30-Second Arm Curl Test | Baseline of the study
  This test is performed with dumbbells. A 2.5-kilogram (5-pound) dumbbell is used for women and a 4-kilogram (8-pound) dumbbell for men. The test is performed in a sitting position. Patients are asked to repeat forearm flexion-supination and extension-pronation movements with the dumbbells in their hands as fast as they can for 30 seconds. The number of moves completed gives the total score.
Weight Lifting Test | Baseline of the study (Assessor 2)
  This test is performed using dumbbells. Reference weights for women are 7 kg and for men are 10 kg. Patients will perform the test with each arm separately. The number of repetitions they can achieve is recorded. The test is performed standing.

SECONDARY OUTCOMES:
Demographic Data Form | Baseline of the study
  This form was created by researchers and it consist of personal informations such as gender, age, body mass index, education, duration of disease, Unified Parkinson's Disease Rating Scale, Modified Hoehn & Yahr stage, using medicine, manual shoulder muscle strength

CONTACTS AND LOCATIONS:
Overall Officials: Murat Emirzeoğlu, PhD, Study Chair — Karadeniz Technical University; Adem Aktürk, PhD, Study Chair — İstanbul Gelişim University; Tuğba Eyigürbüz, PhD, Study Chair — Bağcılar Education and Research Hospital
Locations (1):
- İstanbul Medilife Beylikdüzü Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided